## Participant Consent Form

## Efficacy of pressure pad vs pressure bandage immobilisation for snake bite first aid

Thank you for agreeing to participate in this project which is examining the efficacy of current first aid techniques for snake bite.

| By signing this form you are declaring tha | t you: |
|---|---|
| <ul><li>[] Do NOT have a known allergy to venom)</li></ul> | Technetium-99m sulfur colloid (the mock |
| <ul> <li>[] Do NOT have a known or clinical lymphoedema, lymph node surge</li> <li>[] Do NOT have known lymphoma</li> <li>[] Do NOT have known heart failure</li> <li>[] Do NOT have known kidney dise</li> <li>[] Do NOT have known liver diseas</li> <li>[] Do NOT have known peripheral value</li> </ul> | ery etc) e ase e |
| | e able to undertake a series of 6 scans over a<br>ble that will be developed with you after you |
| | nderstand what is required of your participation of provided to you and as the result of any igator team. |
| series you will be given a \$100 gift card in | t upon your completion of the project scan gratitude for your participation and time, and to completion you will be ineligible for this. |
| | t your participation is entirely voluntary and r consent for participation in the project at any |
| 1 | DOB: give my |
| consent to participate in the project nam provided above is correct to the best of m | ed above and declare that all information |
| Signed: | Date: |
| Investigator name: | Signature: |